CLINICAL TRIAL: NCT06754176
Title: Full-Avoidance vs. Permissive/Regulated Drinking & Outcomes On Fibrillation (FULL-PROOF)
Brief Title: Full-Avoidance vs. Permissive/Regulated Drinking & Outcomes On Fibrillation
Acronym: FULL-PROOF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 24-41856; R01AA022222 (NIH)
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation (AF); Atrial Fibrillation (Paroxysmal)
Keywords: Alcohol; Drinking; Mediterranean Drinking Pattern; Atrial Fibrillation; AFib; AF; Heart Rhythm
MeSH Terms: conditions — Atrial Fibrillation | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: This is a randomized, case-crossover trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol Non-Avoidance Case-Crossover Arm (Experimental): On a given day of the 14-day study period, participants may be randomly assigned to not avoid consuming alcohol. All participants will be instructed that any alcohol consumed should not be more than 2 drinks in a 24 hour period for men and not more than 1 drink in a 24 hour period for women.
  The frequency of randomization will be tailored to the baseline usual frequency of alcohol consumption: For example, those who drink an average of 4 days a week/don't drink 3 days a week will have their randomization programmed to assure an average of 7 non-drinking days over the two-week period. Participants will not receive the same randomization assignment more than two consecutive days in a row.
  Participants will press a button on their continuously recording ECG monitor to time-stamp every alcohol drink consumed.
  Interventions: Behavioral: Alcohol Consumption Randomized Instructions
- Alcohol Avoidance Case-Crossover Arm (Experimental): On a given day of the 14-day study period, participants may be randomly assigned to avoid consuming alcohol.
  The frequency of randomization will be tailored to the baseline usual frequency of alcohol consumption: For example, those who drink an average of 4 days a week/don't drink 3 days a week will have their randomization programmed to assure an average of 7 non-drinking days over the two-week period. Participants will not receive the same randomization assignment more than two consecutive days in a row.
  Interventions: Behavioral: Alcohol Consumption Randomized Instructions

INTERVENTIONS:
Behavioral: Alcohol Consumption Randomized Instructions — Alcohol Avoidance: In this intervention assignment, participants will be instructed to avoid drinking alcohol for this day.
  Alcohol Non-Avoidance: In this intervention assignment, participants will be allowed to drink alcohol for this day.

SUMMARY:
The goal of this study is to assess the short-term effects of minimal and moderate drinking on atrial fibrillation (AFib) episodes in a real-world population diagnosed with 'come-and-go'/paroxysmal AFib. The question it aims to answer is:

Is there a greater occurrence of AFib episodes when participants are allowed to consume alcohol according to random assignment?

Participants will:

* Be given daily random assignments to avoid or not to avoid alcohol
* Wear an adhesive electrocardiographic (ECG) heart monitor
* Wear a wrist-worn fitness tracker
* Wear an anklet transdermal alcohol monitor
* Wear an adhesive glucose monitor
* Complete morning and evening surveys daily

Participants may be compensated up to $50 for full completion of the study. This study can be done in-person or remote.

DETAILED DESCRIPTION:
This study is a case-crossover randomized trial, where each participant will be instructed to avoid or not avoid drinking alcohol on randomly assigned days during a 14-day monitoring period. Participants will also wear an external ECG monitor, an alcohol monitor, a continuous glucose monitor, and a fitness tracker for up to two weeks while utilizing a mobile application to receive daily instructions/reminders on drinking and short surveys. The investigators will compare participant self-report of alcohol consumption, glucose monitoring, fitness levels, sleep health, and heart rhythm data in order to better understand the immediate relationship between drinking alcohol and heart rhythm. A total of 100 participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria

* Comfortable reading and writing in English
* Have a smartphone and willing and able to use the Eureka mobile application
* Currently diagnosed with paroxysmal AFib without a plan to change their AFib management during the two-week monitoring period
* At least one episode of AFib in the past month OR, in the judgement of a healthcare provider, could potentially have one episode of AF in the next month
* Drank alcohol at least 1 day/week on average in the past month
* Willing and able to be randomly assigned daily to avoid or not avoid drinking alcohol over a 2-week period
* Willing and able to provide written informed consent

Exclusion Criteria

* Only post-operative AFib
* Greater than 40% ventricular pacing
* History of alcohol addiction or abuse determined by self-reported history or AUDIT-C score
* Intolerance to alcohol
* History of liver disease
* Currently incarcerated
* Currently pregnant or trying to get pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Presence or Absence of Discrete Atrial Fibrillation Episodes | 2 weeks
  Participants will be wearing a continuously recording ECG monitor for two weeks. The primary outcome will be the presence (versus absence) of at least one AFib episode on randomly assigned drinking versus non-drinking days.

SECONDARY OUTCOMES:
As-Treated Relationships versus the Presence of AFib | 2 weeks
  As-treated (whether alcohol was consumed or not according to real-time patient reports using the Zio patch button and/ or alcohol sensors) relationships versus the presence of AFib will be considered.
Daily Glucose Levels | 2 weeks
  This will first be assessed according to intention-to-treat and then as-treated. Participants will be wearing a continuous glucose monitor that will record serum glucose levels. A secondary outcome will be difference in daily glucose levels due to alcohol consumption or avoidance during the monitoring period.
Step Counts | 2 weeks
  This will first be assessed according to intention-to-treat and then as-treated. Participants will be wearing a fitness tracker that will record step counts. A secondary outcome will be difference in step counts due to alcohol consumption or avoidance during the monitoring period.
Sleep Duration | 2 weeks
  This will first be assessed according to intention-to-treat and then as-treated. Participants will be wearing a fitness tracker that will record sleep duration. A secondary outcome will be difference in sleep duration due to alcohol consumption or avoidance during the monitoring period.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Marcus, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Medical Center at Parnassus, San Francisco, California
  - UCSF Medical Center at Mission Bay, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Al-Khatib SM, Desvigne-Nickens P, Alonso A, Djousse L, Forman DE, Gillis AM, Hendriks JML, Hills MT, Kirchhof P, Link MS, Marcus GM, Mehra R, Murray KT, Parkash R, Pina IL, Redline S, Rienstra M, Sanders P, Somers VK, Van Wagoner DR, Wang PJ, Cooper LS, Go AS. Research Priorities in the Secondary Prevention of Atrial Fibrillation: A National Heart, Lung, and Blood Institute Virtual Workshop Report. J Am Heart Assoc. 2021 Aug 17;10(16):e021566. doi: 10.1161/JAHA.121.021566. Epub 2021 Aug 5. PMID 34351783
- [Background] Chung MK, Eckhardt LL, Chen LY, Ahmed HM, Gopinathannair R, Joglar JA, Noseworthy PA, Pack QR, Sanders P, Trulock KM; American Heart Association Electrocardiography and Arrhythmias Committee and Exercise, Cardiac Rehabilitation, and Secondary Prevention Committee of the Council on Clinical Cardiology; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular and Stroke Nursing; and Council on Lifestyle and Cardiometabolic Health. Lifestyle and Risk Factor Modification for Reduction of Atrial Fibrillation: A Scientific Statement From the American Heart Association. Circulation. 2020 Apr 21;141(16):e750-e772. doi: 10.1161/CIR.0000000000000748. Epub 2020 Mar 9. PMID 32148086
- [Background] Voskoboinik A, Kalman JM, De Silva A, Nicholls T, Costello B, Nanayakkara S, Prabhu S, Stub D, Azzopardi S, Vizi D, Wong G, Nalliah C, Sugumar H, Wong M, Kotschet E, Kaye D, Taylor AJ, Kistler PM. Alcohol Abstinence in Drinkers with Atrial Fibrillation. N Engl J Med. 2020 Jan 2;382(1):20-28. doi: 10.1056/NEJMoa1817591. PMID 31893513
- [Background] Stewart S, Hart CL, Hole DJ, McMurray JJ. Population prevalence, incidence, and predictors of atrial fibrillation in the Renfrew/Paisley study. Heart. 2001 Nov;86(5):516-21. doi: 10.1136/heart.86.5.516. PMID 11602543
- [Background] Mukamal KJ, Tolstrup JS, Friberg J, Jensen G, Gronbaek M. Alcohol consumption and risk of atrial fibrillation in men and women: the Copenhagen City Heart Study. Circulation. 2005 Sep 20;112(12):1736-42. doi: 10.1161/CIRCULATIONAHA.105.547844. Epub 2005 Sep 12. PMID 16157768
- [Background] Mukamal KJ, Psaty BM, Rautaharju PM, Furberg CD, Kuller LH, Mittleman MA, Gottdiener JS, Siscovick DS. Alcohol consumption and risk and prognosis of atrial fibrillation among older adults: the Cardiovascular Health Study. Am Heart J. 2007 Feb;153(2):260-6. doi: 10.1016/j.ahj.2006.10.039. PMID 17239687
- [Background] Frost L, Vestergaard P. Alcohol and risk of atrial fibrillation or flutter: a cohort study. Arch Intern Med. 2004 Oct 11;164(18):1993-8. doi: 10.1001/archinte.164.18.1993. PMID 15477433
- [Background] Djousse L, Levy D, Benjamin EJ, Blease SJ, Russ A, Larson MG, Massaro JM, D'Agostino RB, Wolf PA, Ellison RC. Long-term alcohol consumption and the risk of atrial fibrillation in the Framingham Study. Am J Cardiol. 2004 Mar 15;93(6):710-3. doi: 10.1016/j.amjcard.2003.12.004. PMID 15019874
- [Background] Engel TR, Luck JC. Effect of whiskey on atrial vulnerability and "holiday heart". J Am Coll Cardiol. 1983 Mar;1(3):816-8. doi: 10.1016/s0735-1097(83)80195-8. PMID 6826972
- [Background] Lowenstein SR, Gabow PA, Cramer J, Oliva PB, Ratner K. The role of alcohol in new-onset atrial fibrillation. Arch Intern Med. 1983 Oct;143(10):1882-5. PMID 6625772
- [Background] Ettinger PO, Wu CF, De La Cruz C Jr, Weisse AB, Ahmed SS, Regan TJ. Arrhythmias and the "Holiday Heart": alcohol-associated cardiac rhythm disorders. Am Heart J. 1978 May;95(5):555-62. doi: 10.1016/0002-8703(78)90296-x. No abstract available. PMID 636996
- [Background] Koskinen P, Kupari M, Leinonen H, Luomanmaki K. Alcohol and new onset atrial fibrillation: a case-control study of a current series. Br Heart J. 1987 May;57(5):468-73. doi: 10.1136/hrt.57.5.468. PMID 3593617
- [Background] Marcus GM, Dukes JW, Vittinghoff E, Nah G, Badhwar N, Moss JD, Lee RJ, Lee BK, Tseng ZH, Walters TE, Vedantham V, Gladstone R, Fan S, Lee E, Fang C, Ogomori K, Hue T, Olgin JE, Scheinman MM, Hsia H, Ramchandani VA, Gerstenfeld EP. A Randomized, Double-Blind, Placebo-Controlled Trial of Intravenous Alcohol to Assess Changes in Atrial Electrophysiology. JACC Clin Electrophysiol. 2021 May;7(5):662-670. doi: 10.1016/j.jacep.2020.11.026. Epub 2021 Jan 27. PMID 33516710
- [Background] Aung S, Nah G, Vittinghoff E, Groh CA, Fang CD, Marcus GM. Population-Level Analyses of Alcohol Consumption as a Predictor of Acute Atrial Fibrillation Episodes. Nat Cardiovasc Res. 2022 Jan;1(1):23-27. doi: 10.1038/s44161-021-00003-7. Epub 2022 Jan 12. No abstract available. PMID 38037649
- [Background] McManus DD, Yin X, Gladstone R, Vittinghoff E, Vasan RS, Larson MG, Benjamin EJ, Marcus GM. Alcohol Consumption, Left Atrial Diameter, and Atrial Fibrillation. J Am Heart Assoc. 2016 Sep 14;5(9):e004060. doi: 10.1161/JAHA.116.004060. PMID 27628571
- [Background] Mandyam MC, Vedantham V, Scheinman MM, Tseng ZH, Badhwar N, Lee BK, Lee RJ, Gerstenfeld EP, Olgin JE, Marcus GM. Alcohol and vagal tone as triggers for paroxysmal atrial fibrillation. Am J Cardiol. 2012 Aug 1;110(3):364-8. doi: 10.1016/j.amjcard.2012.03.033. Epub 2012 Apr 20. PMID 22521307
- [Background] Dukes JW, Dewland TA, Vittinghoff E, Olgin JE, Pletcher MJ, Hahn JA, Gladstone RA, Marcus GM. Access to alcohol and heart disease among patients in hospital: observational cohort study using differences in alcohol sales laws. BMJ. 2016 Jun 14;353:i2714. doi: 10.1136/bmj.i2714. PMID 27301557
- [Background] Whitman IR, Agarwal V, Nah G, Dukes JW, Vittinghoff E, Dewland TA, Marcus GM. Alcohol Abuse and Cardiac Disease. J Am Coll Cardiol. 2017 Jan 3;69(1):13-24. doi: 10.1016/j.jacc.2016.10.048. PMID 28057245
- [Background] Marcus GM, Smith LM, Whiteman D, Tseng ZH, Badhwar N, Lee BK, Lee RJ, Scheinman MM, Olgin JE. Alcohol intake is significantly associated with atrial flutter in patients under 60 years of age and a shorter right atrial effective refractory period. Pacing Clin Electrophysiol. 2008 Mar;31(3):266-72. doi: 10.1111/j.1540-8159.2008.00985.x. PMID 18307620
- [Background] Groh CA, Faulkner M, Getabecha S, Taffe V, Nah G, Sigona K, McCall D, Hills MT, Sciarappa K, Pletcher MJ, Olgin JE, Marcus GM. Patient-reported triggers of paroxysmal atrial fibrillation. Heart Rhythm. 2019 Jul;16(7):996-1002. doi: 10.1016/j.hrthm.2019.01.027. Epub 2019 Feb 14. PMID 30772533
- [Background] Marcus GM, Modrow MF, Schmid CH, Sigona K, Nah G, Yang J, Chu TC, Joyce S, Gettabecha S, Ogomori K, Yang V, Butcher X, Hills MT, McCall D, Sciarappa K, Sim I, Pletcher MJ, Olgin JE. Individualized Studies of Triggers of Paroxysmal Atrial Fibrillation: The I-STOP-AFib Randomized Clinical Trial. JAMA Cardiol. 2022 Feb 1;7(2):167-174. doi: 10.1001/jamacardio.2021.5010. PMID 34775507
- [Background] Marcus GM, Vittinghoff E, Whitman IR, Joyce S, Yang V, Nah G, Gerstenfeld EP, Moss JD, Lee RJ, Lee BK, Tseng ZH, Vedantham V, Olgin JE, Scheinman MM, Hsia H, Gladstone R, Fan S, Lee E, Fang C, Ogomori K, Fatch R, Hahn JA. Acute Consumption of Alcohol and Discrete Atrial Fibrillation Events. Ann Intern Med. 2021 Nov;174(11):1503-1509. doi: 10.7326/M21-0228. Epub 2021 Aug 31. PMID 34461028